CLINICAL TRIAL: NCT05890222
Title: IMPlementation of Evidence Based Facility and Community Interventions to Reduce the Treatment Gap for depRESSion
Acronym: IMPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Harvard Medical School (HMS and HSDM) (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAN_IMPRESS_2023
Record Dates: First submitted 2023-05-12; First posted 2023-06-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Model (Experimental): In addition to the facility model, village clusters in this arm will receive community intervention strategies delivered by community volunteers.
  Interventions: Behavioral: Community Intervention; Behavioral: Healthy Activity Program (HAP)
- Facility Model (Active Comparator): The HAP, a manualized and evidence-based psychological treatment based on behavioural activation, will be delivered by existing healthcare workers (called counsellors from here onwards) within the health centres who will be trained to deliver the HAP.
  Interventions: Behavioral: Healthy Activity Program (HAP)

INTERVENTIONS:
Behavioral: Community Intervention — Community intervention strategies will be delivered by community volunteers (called Sangathis - which means companion in Konkani, one of the local languages) to i) enhance demand for the HAP treatment and ii) promote engagement with, and completion of, the HAP treatment. The community intervention is co-produced with local community members and includes strategies such as activities to increase awareness about depression (community meetings, street plays and health camps), and dissemination of psycho-educational materials (i.e., leaflets and posters), identify people with possible depression in the community, and facilitate access to HAP in the health centres. Additionally, the Sangathis will coordinate continuing care of people receiving HAP, through home visits to encourage behavioural activation, homework completion and following up with the counsellor, and engaging family members to support the patient in achieving treatment goals.
  Arms: Community Model
Behavioral: Healthy Activity Program (HAP) — HAP includes the following strategies: psychoeducation, behavioural assessment, activity monitoring, activity structuring and scheduling, activation of social networks, and problem-solving. HAP will be delivered in an individual format. It entails three phases of treatment, delivered over six to eight sessions, each lasting up to 40 minutes, with the sessions being at weekly intervals. Sessions will be delivered face-to-face, at the health centre where the counsellors already work.

SUMMARY:
The goal of this Hybrid Type 2 Implementation-Effectiveness Cluster Randomised Controlled Trial is to reduce the treatment gap for depression through the integrated implementation of interventions in facility and community platforms, in Goa, India. The primary question is to examine whether a community intervention ("Community Model") enhances the demand for, and improves the outcomes of, an evidence-based, brief psychological treatment for depression delivered by non-specialist health workers in primary health care facilities ("Facility Model"). Participants in the Facility Model arm will receive only a psychosocial intervention for depression (the Healthy Activity Program - HAP) while participants in the Community Model will receive both the HAP and the community intervention. We will compare the Facility Model and the Community Model to assess if the latter is superior in increasing the demand for depression treatment in primary care, increasing uptake of treatment by people with depression, increasing treatment completion rates, and reducing the severity of depression.

ELIGIBILITY:
(A) Contact Coverage Outcome

Inclusion Criteria

* Adults (>18 years)
* Residing in the clusters included in the trial
* Speak English or one of the local languages (Konkani, Marathi, Hindi)

Exclusion Criteria

* Patients with significant speech, hearing, or language impairment that interferes with completion of the screening and/or receipt of psychosocial intervention
* Patients who present to the health centre for emergency medical attention
* Patients with active psychotic symptoms

(B) Effectiveness Coverage Outcome

Inclusion Criteria

* Adults (>18 years);
* Residing in the clusters included in the trial
* Speak English or one of the local languages (Konkani, Marathi, Hindi).
* Screen positive for moderately severe or severe depression (total score >14) on the Patient Health Questionnaire-9 items (PHQ-9)

Exclusion Criteria

* Patients with significant speech, hearing, or language impairment that interferes with completion of the screening and/or receipt of psychosocial intervention
* Patients who present to the health centre for emergency medical attention
* Patients with active psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Contact coverage | During recruitment
  Patient Health Questionnaire 9 items (PHQ-9) score >4. The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.
Effectiveness coverage | Three months post recruitment
  Mean Patient Health Questionnaire 9 items (PHQ-9 score). The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Sustained effectiveness | Six months post recruitment
  Mean Patient Health Questionnaire 9 items (PHQ-9 score). The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.
Remission | Three months post recruitment
  Patient Health Questionnaire 9 items (PHQ-9 score) score <10. . The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.
Remission | Six months post recruitment
  Patient Health Questionnaire 9 items (PHQ-9 score) score <10. . The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.
Response to treatment | Three months post recruitment
  >50% reduction in Patient Health Questionnaire 9 items (PHQ-9 score) score. The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.
Response to treatment | Six months post recruitment
  >50% reduction in Patient Health Questionnaire 9 items (PHQ-9 score) score. The minimum score is 0 and maximum score is 27; with higher scores indicating greater severity of depression.
Client Service Receipt Inventory | 3- and 6- months post recruitment
  Out-of-pocket costs for receiving care and the related non-medical costs
WHO Disability Assessment Schedule (WHODAS 2.0) | Baseline, 3- and 6- months post recruitment
  Standardized disability scores used to estimate Quality Adjusted Life Years (QALYs). The 12-item WHODAS 2.0 score ranges from 12 to 60, where higher scores indicate higher disability or loss of function.
Survey form for collecting costs of receiving HAP intervention to patients | 3 months post recruitment
  Out-of-pocket costs for receiving HAP intervention (e.g. time loss, travel)
Inventory form for collecting system-level economic costs of delivering interventions | Monthly, through study completion up to approximately 12 months
  System-level costs: Economic costs in WHO six building blocks for delivering the interventions
Depression awareness | Baseline, 6, 12 and 18 months of implementation
  Awareness about depression. This will be a bespoke tool developed for our trial and will have questions to assess awareness related to depression based on the information disseminated in our community intervention and higher scores will indicate greater awareness.
Perceived social support | 3- and 6- months post recruitment
  Perception of social support received. This will be a bespoke tool developed for our trial and will have questions to assess perceived support related to support provided by community volunteers in our community intervention and higher scores will indicate greater support.
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, 3- and 6-months post-recruitment
  12 item short instrument designed to measure an individual's perception of support from 3 sources: family, friends and a significant other. Minimum score 12 and maximum 84
Treatment completion | Across 12 months of implementation
  Met treatment goals or completed the maximum number of sessions or were referred to mental health specialists
Behavioral activation | Baseline, 3- and 6- months post recruitment.
  Level of behavioral activation measured using PREMIUM Abbreviated Activation Scale. This is a five-item scale, originally developed based on the Behavioural Activation for Depression Scale. It includes five self-reported indicators and the total score can range from 0 to 20. Higher scores indicate greater level of behavioural activation such as engagement with a variety of activities, and associated pleasure and mastery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sangath, Mormugao, Goa, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nadkarni A, Gandhi Y, Fernandes L, Mirchandani K, Kamat S, Weiss HA, Singla DR, Velleman R, Lu C, Bhatia U, Biswal B, Sequeira M, D'souza E, Raikar K, Patel V. Effectiveness and cost-effectiveness of a community intervention in enhancing access to care and improving clinical outcomes for depression: a protocol for a cluster randomised controlled trial in India. Trials. 2024 Aug 28;25(1):569. doi: 10.1186/s13063-024-08236-0. PMID 39198915